CLINICAL TRIAL: NCT00328055
Title: Effects of an Easy to Read Advance Directive on Acceptability, Knowledge, and Self-efficacy Compared to a Standard Advance Directive
Brief Title: Comparison of an Easy to Read Advance Directive Versus a Standard Advance Directive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: AG0066; 5T32AG000212-14 (NIH); 5K07AG000912-05 (NIH); 5R01AG023626-02 (NIH); 5K23RR016539-05 (NIH)
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Aging
Keywords: functional ability; patient care management; communication; literacy
MeSH Terms: conditions — Communication; Literacy

INTERVENTIONS:
Behavioral: AD-Easy (Advance Directive-Easy)
Behavioral: AD-Standard (Advance Directive-Standard)

SUMMARY:
The purpose of this study is to compare the acceptability, usefulness, self-efficacy and comprehension of an easy-to-read advance directive form versus a standard advance directive form written at a post graduate reading level.

DETAILED DESCRIPTION:
Advance directives are forms that allow patients to document their medical treatment preferences and to designate another person to help make medical decisions if they were to become too sick to make their own decisions. Most patients, even seriously ill older adults, do not fill out advance directive forms. Since the mean reading level in the US is at the 8th grade level (5th grade for elders) and since most advance directive documents are written beyond a 12th grade reading level, many patients may not be able to read, much less complete, the standard advance directive forms.

This study hypothesized that an advance directive form written at a 5th grade reading level (AD-Easy) that included culturally appropriate graphics explaining the text, and also included questions concerning patients' values, would be preferred over the standard advance directive form being used in California (AD-Standard).

The participant's literacy level and baseline knowledge of advance directive topics were assessed. Participants were then stratified by literacy level to be randomized to first attempt to read and complete either the AD-Easy or the AD-Standard. Then the participant's acceptance of the forms, self-efficacy or confidence with treatment decisions, attitudes about the form's utility, and post form review comprehension were assessed. Participants then crossed over to review the alternate form and were asked to state which form they preferred to take home. Six months later participants were called and asked if they had thought about their medical treatment preferences, spoken to their family, friends, or doctor about their treatment preferences, or if they filled out the advance directive form.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years
* Primary physician in the General Medicine Clinic at San Francisco General Hospital, San Francisco, CA
* English- or Spanish-speaking

Exclusion Criteria:

* Blind
* Deaf
* Delirious
* Demented

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-08; Study Completion 2005-07

PRIMARY OUTCOMES:
Acceptability
self-efficacy
attitudes about the forms utility
comprehension
preference

SECONDARY OUTCOMES:
6 month outcomes included whether participant talked with their doctor about treatment wishes, talked to family, thought about treatment decisions, or filled out an advance directive

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sudore, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Emanuel LL, Barry MJ, Stoeckle JD, Ettelson LM, Emanuel EJ. Advance directives for medical care--a case for greater use. N Engl J Med. 1991 Mar 28;324(13):889-95. doi: 10.1056/NEJM199103283241305. PMID 2000111
- [Background] Ott BB, Hardie TL. Readability of advance directive documents. Image J Nurs Sch. 1997 Spring;29(1):53-7. doi: 10.1111/j.1547-5069.1997.tb01140.x. PMID 9127541
- [Background] Nolan MT. Could lack of clarity in written advance directives contribute to their ineffectiveness? A study of the content of written advance directives. Appl Nurs Res. 2003 Feb;16(1):65-9. doi: 10.1053/apnr.2003.50007. PMID 12624865
- [Background] Jacobson TA, Thomas DM, Morton FJ, Offutt G, Shevlin J, Ray S. Use of a low-literacy patient education tool to enhance pneumococcal vaccination rates. A randomized controlled trial. JAMA. 1999 Aug 18;282(7):646-50. doi: 10.1001/jama.282.7.646. PMID 10517717
- [Background] Kirsch IS, Jungeblut A, Jenkins L, Kolstad A. Adult Literacy in America: A First Look at the Findings of the National Adult Literacy Survey. Washington, DC: Office of Educational Research and Improvement U.S. Department of Education; 1993 http://nces.ed.gov/pubs93/93275.pdf.